CLINICAL TRIAL: NCT07317895
Title: Sensitivity to Ovarian Hormones and Depression in Adolescents
Acronym: SOHDA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Whitney Hindmarch, Research Manager, University of Calgary
Other Study IDs: REB25-1647
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Depressed
Keywords: Depression; Estrogen; Progesterone
MeSH Terms: conditions — Consciousness Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SOHDA corort: Main study cohort

SUMMARY:
The goal of this observational study is to learn about the relationship between changes in ovarian hormones (estrogen and progesterone) and adolescent depression. The main question it aims to answer is:

Can we identify a subset adolescents assigned female at birth with a history of depression who are particularly sensitive to changes in ovarian hormones? Participants will be monitoring daily absolute ovarian hormone levels at home using the Mira Analyzer and answer online survey questions about their mental health for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth, at least 1 year post-menarche, naturally cycling, history of depression or symptoms of depression, and able to read and write in English.

Exclusion Criteria:

* Pregnant or taking any hormonal or cycle altering medications/devices.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Depressed, naturally cycling adolescents assigned female at birth.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Identification ovarian hormone affect sensitivity | 90 days
  Identify depressed adolescents assigned female at birth with depressed affect sensitivity to changes in ovarian hormones across the menstrual cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No